CLINICAL TRIAL: NCT07287982
Title: A Phase 2 Double-Blinded, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of Intravenous Administration of ARGX-119 in Pediatric Participants Aged 5 to Less Than 18 Years With Spinal Muscular Atrophy
Brief Title: A Study to Assess the Safety, Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of Intravenous Administration of ARGX-119 in Pediatric Participants Aged 5 to Less Than 18 Years With Spinal Muscular Atrophy
Acronym: Sparkle
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARGX-119-24-SMA-2001; 2025-523496-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: Spinal Muscular Atrophy; Pediatric; Muscle Function; Fatigability; SMA; ambulant
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DBTP - ARGX-119 IV (Experimental): Participants receive ARGX-119 IV during the DBTP
  Interventions: Biological: ARGX-119 IV
- DBTP - Placebo IV (Placebo Comparator): Participants receive placebo IV during the DBTP
  Interventions: Other: Placebo IV
- ATEP - ARGX-119 IV (Placebo Comparator): Participants receive ARGX-119 IV during the ATEP. Participants from ARGX-119 IV arm in the DBTP will receive placebo once to maintain the DBTP blinding
  Interventions: Biological: ARGX-119 IV; Other: Placebo IV

INTERVENTIONS:
Biological: ARGX-119 IV — Intravenous infusion of ARGX-119
  Arms: ATEP - ARGX-119 IV; DBTP - ARGX-119 IV
Other: Placebo IV — Intravenous infusion of placebo
  Arms: ATEP - ARGX-119 IV; DBTP - Placebo IV

SUMMARY:
This study aims to find the correct dose of ARGX-119 for children with SMA. The study will also look at how safe the study drug is, how well it works, how it moves through the body, and how the immune system responds to it. The study consists of a double-blinded treatment period (DBTP) where participants will either receive ARGX-119 IV or placebo IV, in addition to disease-modifying therapy (DMT) for 24 weeks. Participants who complete the DBTP will enter the open-label active-treatment extension period (ATEP) during which all participants will receive ARGX-119 IV up to 100 weeks (approximately 2 years).

DETAILED DESCRIPTION:
This phase 2 study aims to establish proof of concept with the age-appropriate dose of ARGX-119 in ambulant pediatric patients with spinal muscular atrophy (SMA). Despite available treatments, there remains an unmet medical need for patients with SMA. Neuromuscular junction (NMJ) dysfunction contributes to the pathophysiology of SMA, including muscle weakness and fatigability. Activation of muscle-specific kinase (MuSK) by ARGX-119 may stabilize and improve NMJ function in patients with SMA, reducing muscle weakness and fatigability, and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Is aged ≥5 to <18 years when completing the informed consent process, defined as providing informed assent according to local regulations and having a parent or guardian sign the ICF, and can comply with protocol
* requirements.
* Has documented historical genetic diagnosis of 5q-SMA.
* Currently receiving a stable SMA treatment regimen (nusinersen or risdiplam) and/or have a history of onasemnogene abeparvovec treatment
* Must be able to walk at least 50 meters without walking aids in the 6MWT at screening

Exclusion Criteria:

* Known medical condition that would interfere with an accurate assessment of SMA, confound the results of the study, or put the participant at undue risk, as assessed by the investigator
* Recent major surgery, except spinal fusion, within 3 months of screening or intends to have major surgery during the study
* Current or previous administration of antimyostatin therapies in the past 6 months
* Severe scoliosis (defined as curvature >40°) and/or contractures at screening. o History of spinal fusion within 6 months before screening or planned during the study
* Respiratory insufficiency, defined by the medical necessity for invasive or noninvasive ventilation for daytime treatment while awake. Ventilation used overnight or during daytime naps is acceptable.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2029-05-28 (Estimated); Study Completion 2029-05-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | Up to 124 weeks
  Adverse Events
Incidence of SAEs | Up to 124 weeks
  Serious Adverse Events
Change in RHS total score from baseline to week 24 of the double blinded treatment period (DBTP) | Up to 24 weeks
  The RHS (Revised Hammersmith Scale) is a validated 36-item scale developed to evaluate the spectrum of gross motor function. Maximum total score; 69 (optimal motor function)

SECONDARY OUTCOMES:
Change from baseline over time for the 6MWT - distance and fatigue index | Up to 124 weeks
  In the 6MWT (6-minute walk test) participants will be instructed to walk as fast as possible without jogging or running along a 25- meter linearly marked course for 6 minutes without using walking devices or assistance. Distance walked over the entire 6-minute period, and other parameters, will be determined
ARGX-119 serum concentrations over time | Up to 124 weeks
  ARGX-119 serum concentrations over time
Incidence of antidrug antibodies (ADA) against ARGX-119 | Up to 124 weeks
  Incidence of antidrug antibodies (ADA) against ARGX-119

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Childrens Hospital, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Rare Disease Research FL LLC, Kissimmee, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - Rare Disease Research NC, LLC, Hillsborough, North Carolina
  - Children's Hospital Philadelphia - Neurology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Neurology Rare Disease Center, Flower Mound, Texas
  - Texas Children's Hospital, Houston, Texas
  - Childrens Hospital of The Kings Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No